CLINICAL TRIAL: NCT01751802
Title: An Outpatient Phase 3 Efficacy Study of Ecopipam (PSYRX 101) in the Symptomatic Treatment of Self-Injurious Behavior in Subjects With Lesch-Nyhan Disease
Brief Title: Ecopipam Treatment of Self-Injurious Behavior in Subjects With Lesch-Nyhan Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated for commercial reasons
Sponsor: Emalex Biosciences Inc. (Industry)
Collaborators: Psyadon Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PSY102
Record Dates: First submitted 2012-12-14; First posted 2012-12-18 (Estimated); Results first posted 2015-10-08 (Estimated); Last update posted 2024-04-22 (Actual); Status verified 2015-10

CONDITIONS: Lesch-Nyhan Disease; Self-injurious Behavior
Keywords: Lesch Nyhan Disease; Self-Injury
MeSH Terms: conditions — Lesch-Nyhan Syndrome; Self-Injurious Behavior | interventions — ecopipam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ecopipam (Experimental): Active substance being tested, orally once a day at bedtime
  Interventions: Drug: Ecopipam
- Placebo (Placebo Comparator): Inactive substance being tested, orally once a day at bedtime
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ecopipam — Antagonist of the dopamine D1 receptor
  Other Names: PSYRX 101; SCH 39166
  Arms: Ecopipam
Drug: Placebo — Placebo for Ecopipam
  Arms: Placebo

SUMMARY:
The purpose of this research study is to gather scientific information about the effectiveness and safety of the study drug, Ecopipam (PSYRX 101), for the treatment of self-injurious behaviors when compared with the effectiveness and safety of placebo (inactive substance) in subjects with Lesch-Nyhan Disease.

DETAILED DESCRIPTION:
This study will be done in approximately 6 centers in approximately 4 countries, and approximately 24 subjects will be included. This study is divided into two parts. The first is a double-blinded portion lasting up to 18 weeks in total. The second portion is an optional open-label extension and lasts up to 54 weeks total. The total duration of the study, if you choose to participate in both portions, is anticipated to be up to approximately 78 weeks.

The first portion of this study is double-blind and assignment to a treatment group is done randomly. In this study, there are two treatment groups. One group will receive Ecopipam for one 6-week period and placebo for two 6-week periods, and the other group will receive Ecopipam for two 6-week periods and placebo for one 6-week period.

Subjects who did not experience any clinically significant side effects during the blinded portion of the study may be eligible to participate in an open-label extension that may last up to 54 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have classic LND as defined by (a) characteristic clinical syndrome (evidence of overproduction of uric acid, severe generalized dystonia, frequent and persistent self-injurious behavior (SIB), and cognitive impairment) and (b) laboratory confirmation for mutation of the HPRT gene or severe deficiency of the associated enzyme.
* Subjects must have a minimum combined score of 20 on the Behavior Problems Inventory (BPI) SIB subscales for frequency and severity as assessed by the caregiver.
* Subjects must have a minimum score of 4 on the Physician's Global Impression (PGI) severity scale.
* Subject must be ≥ 6 years old.
* Subjects must weigh > 10 kg.

Exclusion Criteria:

* Subjects who are currently treated with medications for seizures.
* Subjects who are on neuroleptics or dopamine-depleting agents.
* Subjects with impaired renal function as defined by a serum creatinine >1.5 mg/dL.

Ages: 6 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-12; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: H J Jinnah, MD, Principal Investigator — Emory University
Locations (2):
- H.J. Jinnah, Atlanta, Georgia, United States
- Hospital Universitario La Paz, Madrid, Spain

REFERENCES:
- See also: Sponsor's website — http://www.psyadonrx.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Ecopipam Then Placebo Then Ecopipam: Ecopipam, the active substance being tested, 100mg tablets for body weight > 20kg OR 50 mg tablets for body weight up to 20kg, once daily at bedtime for 6 weeks; then Placebo, the inactive substance being tested to be taken once a day at bedtime for 6 weeks; then Ecopipam, the active substance being tested, 100mg tablets for body weight > 20kg OR 50 mg tablets for body weight up to 20kg, once daily at bedtime for 6 weeks
- Placebo Then Ecopipam Then Placebo: Placebo, the inactive substance being tested to be taken once a day at bedtime for 6 weeks; then Ecopipam, the active substance being tested, 100mg tablets for body weight > 20kg OR 50 mg tablets for body weight up to 20kg, once daily at bedtime for 6 weeks; then Placebo, the inactive substance being tested to be taken once a day at bedtime for 6 weeks
Period: Overall Study
Arm/Group | Ecopipam Then Placebo Then Ecopipam | Placebo Then Ecopipam Then Placebo
Started | 5 | 4
Completed Period 1 | 2 | 4
Completed Period 2 | 2 | 1
Completed Period 3 | 2 | 1
Completed | 1 | 2
Not Completed | 4 | 2
Not completed — Adverse Event | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ecopipam Then Placebo Then Ecopipam | Placebo Then Ecopipam Then Placebo | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Continuous [Mean (Full Range); unit: years] | 10.8 [6 to 22] | 9.8 [6 to 12] | 10.3 [6 to 22]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 5 | 4 | 9
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 3
  Spain | 3 | 3 | 6
Weight [Mean (Full Range); unit: kg] | 28.3 [16.5 to 55.4] | 21.9 [16.0 to 26.5] | 25.4 [16.0 to 55.4]
BMI [Mean (Full Range); unit: kg/m^2] | 15.6 [13.9 to 18.1] | 13.8 [13.1 to 15.5] | 14.8 [13.1 to 18.1]

OUTCOME MEASURES:

1. Primary Outcome: Behavior Problems Inventory - Self-Injurious Behavior Subscale
Description: The primary endpoint is the BPI (SIB subscales - total for frequency and severity) as assessed by the caregiver. BPI Self-Injurious Behavior Subscale ranges from 0 to 45, with higher scores indicating more self-injurious behavior.
Time Frame: Baseline, end of period 1 (6 weeks), end of period 2 (12 weeks), end of period 3 (18 weeks),
Population: All participants who completed the BPI-Self Injurious Behavior survey for 3 or more time points
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Subject #1: Ecopipam Then Placebo Then Ecopipam; Subject #2: Ecopipam Then Placebo Then Ecopipam: Ecopipam, the active substance being tested, 100mg tablets for body weight > 20kg OR 50 mg tablets for body weight up to 20kg, once daily at bedtime for 6 weeks; then Placebo, the inactive substance being tested to be taken once a day at bedtime for 6 weeks; then Ecopipam, the active substance being tested, 100mg tablets for body weight > 20kg OR 50 mg tablets for body weight up to 20kg, once daily at bedtime for 6 weeks
- Subject #3: Placebo Then Ecopipam Then Placebo; Subject #4: Placebo Then Ecopipam Then Placebo: Placebo, the inactive substance being tested to be taken once a day at bedtime for 6 weeks; then Ecopipam, the active substance being tested, 100mg tablets for body weight > 20kg OR 50 mg tablets for body weight up to 20kg, once daily at bedtime for 6 weeks; then Placebo, the inactive substance being tested to be taken once a day at bedtime for 6 weeks
Arm/Group | Subject #1: Ecopipam Then Placebo Then Ecopipam | Subject #2: Ecopipam Then Placebo Then Ecopipam | Subject #3: Placebo Then Ecopipam Then Placebo | Subject #4: Placebo Then Ecopipam Then Placebo
Number analyzed (Participants) | 1 | 1 | 1 | 1
scores on a scale
  BPI Self-Injurious Behavior Subscale, Baseline | 26 | 10 | 78 | 27
  BPI Self-Injurious Behavior Subscale, 6 weeks | 24.1 | 4.3 | 58.3 | 22.6
  BPI Self-Injurious Behavior Subscale, 12 weeks | 25.2 | 11.6 | 21.5 | 16.0
  BPI Self-Injurious Behavior Subscale, 18 weeks | 21 | 6.6 | 28.7 | NA — participant did not complete subscale survey at 18 wks

2. Secondary Outcome: Effect of Ecopipam Withdrawal and Maintenance
Description: The secondary objectives of this study are to assess the effect of withdrawal and maintenance of ecopipam's effects in subjects with LND. Measured by the number of participants whose score changes significantly from baseline on ecopipam or placebo
Time Frame: Baseline, 6 weeks, 12 weeks, 18 weeks
Population: 0 participants analyzed because data are not reliable
Arm/Group | Ecopipam | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Safety Summary of Ecopipam in Patients With Lesch-Nyhan Disease: Total Number of Serious and Non-Serious Adverse Events Experienced During 3 Double-blind Crossover Periods
Description: An additional objective of the study is to assess the safety of ecopipam in subjects with LND for up to 52 weeks. Total number of serious and non-serious adverse events experienced by participants while receiving ecopipam or placebo. For additional detail, see Adverse Events
Time Frame: Total duration over which participants recieved double-blind ecopipam or placebo, up to 6 or 12 weeks
Population: All participants who received at least one dose
Measure: Number; unit: adverse events
Groups:
- Ecopipam: Active substance being tested, orally once a day at bedtime for 6 weeks
  Ecopipam: Antagonist of the dopamine D1 receptor
- Placebo: Inactive substance being tested, orally once a day at bedtime for 6 weeks
  Placebo: Placebo for Ecopipam
Arm/Group | Ecopipam | Placebo
Number analyzed (Participants) | 9 | 6
adverse events
  Non-Serious | 42 | 7
  Serious | 2 | 1

ADVERSE EVENTS:
Time Frame: adverse events collected while participants were receiving ecopipam or placebo, either for 1 period (up to 6 weeks) or 2 periods (up to 12 weeks)
Description: Adverse events were collected for 3 double-blind periods
Arm/Group | Ecopipam | Placebo
Serious Adverse Events (participants affected / at risk) | 2/9 | 1/6
Other Adverse Events (participants affected / at risk) | 8/9 | 2/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ecopipam (N=9) | Placebo (N=6)
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 (1) — During hospitalization, subject also experienced opisthotonus, bronchospasm, hypereosinophilia, & elevated transaminase; all AEs rated as unrelated to ecopipam. Ecopipam continued during hospitalization. All symptoms resolved w/o sequelae.
Dystonic crisis (Nervous system disorders) | 1 | 0 — Subject 05-001 was hospitalized a second time (July 2013) for a dystonic crisis, difficulty swallowing (dysphagia), and depressed mood.
Unusual somnolence (Psychiatric disorders) | 1 | 0 — Subject hospitalized for dysphagia, unusual somnolence and depressed mood, as reported by parents. Causality was rated Reasonable Possibility by investigator. Subject was discharged as somnolence resolved; and subject withdrew because of these AEs.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ecopipam (N=9) | Placebo (N=6)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Agitation (Psychiatric disorders) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Body temperature increased (Investigations) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Compulsive lip biting (Psychiatric disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 3 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 5 (5) | 0 (0)
Dyskinesia (Nervous system disorders) | 0 (0) | 1 (1)
Dystonia (Nervous system disorders) | 2 (2) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1)
Lip injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Opisthotonus (Nervous system disorders) | 2 (2) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Self injurious behaviour (Psychiatric disorders) | 4 (4) | 1 (1)
Somnolence (Nervous system disorders) | 5 (5) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No